CLINICAL TRIAL: NCT01900106
Title: A Prospective, Open-label Trial of Two Abacavir/Lamivudine Based Regimen (ABC/3TC + Darunavir/Ritonavir or ABC/3TC + Raltegravir) in Late Presenter naïve Patients (With CD4 Count <200 Cells/µL - Advanced HIV Disease)
Brief Title: A Prospective, Open-label Trial of Two ABC/3TC Based Regimens in Late Presenter naïve Patients (CD4 <200 Cells/µL)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Modena and Reggio Emilia (Other)
Responsible Party: Principal Investigator, Cristina Mussini, Professor, University of Modena and Reggio Emilia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTLP (PRADAR); 2011-005973-21 (EudraCT Number)
Record Dates: First submitted 2013-07-05; First posted 2013-07-16 (Estimated); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: HIV Infection
Keywords: late presenter; naïve; advanced HIV disease
MeSH Terms: conditions — HIV Infections | interventions — abacavir; Lamivudine; Raltegravir Potassium; abacavir, lamivudine drug combination; Darunavir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- abacavir/lamivudine + raltegravir (Experimental): abacavir/lamivudine + raltegravir
  Interventions: Drug: abacavir/lamivudine + raltegravir
- ABC/3TC + DRV/r (Active Comparator): abacavir/lamivudine + darunavir/ritonavir
  Interventions: Drug: abacavir/lamivudine + darunavir/ritonavir

INTERVENTIONS:
Drug: abacavir/lamivudine + raltegravir — abacavir/lamivudine + raltegravir
  Other Names: Kivexa; Isentress
  Arms: abacavir/lamivudine + raltegravir
Drug: abacavir/lamivudine + darunavir/ritonavir — abacavir/lamivudine + darunavir/ritonavir
  Other Names: Kivexa; Prezista; Norvir
  Arms: ABC/3TC + DRV/r

SUMMARY:
1. PROTOCOL SUMMARY This is a prospective, randomized open-label, 2 arm, 3-phase trial to compare the 48-weeks virological response of two different regimens containing abacavir/lamivudine (abacavir/lamivudine +darunavir/ritonavir (DRV/r) vs abacavir/lamivudine + raltegravir (RAL) in antiretroviral therapy naive, HIV+ individuals presenting for care with CD4+ counts < 200/mm3.

1.1 Clinical Objectives: Primary Objective: To compare the 48-week virological response to two different regimens containing abacavir/lamivudine (abacavir/lamivudine +darunavir/ritonavir (DRV/r) vs abacavir/lamivudine + raltegravir (RAL) in antiretroviral therapy naive, HIV+ individuals presenting for care with CD4+ counts < 200/mm3.

Secondary Objective: a) To compare immunological response at 48 weeks; b) To determine the safety and tolerability of the 2 regimens.

1.2 Study population: 350 in/out patients 1.3 Outcome Primary Endpoint

* Proportion of patients with HIV RNA<50 copies/mL after 48 weeks Secondary Endpoints(s)
* Change in CD4+ cell count from baseline through week 48
* Time to virological rebound 1.4 Study design: Multicentre, parallel group, randomised, open label, non-inferiority study 1.5 Treatment regimens: Arm A: abacavir/lamivudine 1 tablet once a day + raltegravir 400 mg (1 tablet twice a day) Arm B: abacavir/lamivudine 1 tablet once a day + ritonavir 100 mg + darunavir 800 mg once a day.

All drugs have been approved for the treatment of HIV infection. The study population will consist of 350 HIV-positive, HLA B5701-negative patients. At baseline, patients will be randomized 1:1 to start abacavir/lamivudine plus either raltegravir or darunavir/ritonavir. Randomization will be stratified on the basis of the screening CD4+ cell count (≤100 vs ≥100 cells/µL), to ensure balance across treatments groups 1.7 Criteria for Safety: Adverse events and laboratory assessments. 1.8 Statistical analysis: As this is a non-inferiority trial, we will calculate the difference in the proportions of patients experiencing the primary outcome in the two treatment arms and will calculate a 95% confidence interval for this. Non-inferiority of the raltegravir arm will be demonstrated if the lower limit of the 95% confidence interval is greater than -12%. In case non-inferiority will be met, analyses for superiority will be performed.

DETAILED DESCRIPTION:
1. PROTOCOL SUMMARY This is a prospective, randomized open-label, 2 arm, 3-phase trial to compare the 48-weeks virological response of two different regimens containing abacavir/lamivudine (abacavir/lamivudine +darunavir/ritonavir (DRV/r) vs abacavir/lamivudine + raltegravir (RAL) in antiretroviral therapy naive, HIV+ individuals presenting for care with CD4+ counts < 200/mm3.

1.1 Clinical Objectives: Primary Objective: To compare the 48-week virological response to two different regimens containing abacavir/lamivudine (abacavir/lamivudine +darunavir/ritonavir (DRV/r) vs abacavir/lamivudine + raltegravir (RAL) in antiretroviral therapy naive, HIV+ individuals presenting for care with CD4+ counts < 200/mm3.

Secondary Objective:

1. To compare immunological response at 48 weeks;
2. To determine the safety and tolerability of the 2 regimens. 1.2 Study population: 350 inpatients or outpatients will be randomized 1.3 Outcome Primary Endpoint

   * Proportion of patients with undetectable viremia (HIV RNA<50 copies/mL) after 48 weeks Secondary Endpoints(s)
   * Change in CD4+ cell count from baseline through week 48
   * Time to virological rebound Safety endpoints
   * Incidence of adverse events (AEs)
   * Incidence of serious adverse events (SAEs)
   * Discontinuations due to adverse events
   * Incidence of grade 3 or 4 laboratory abnormalities. 1.4 Study design Multicentre, parallel group, randomised, open label, non-inferiority study 1.5 Planned sample size: The planned sample size for this trial is 350 patients 1.6 Treatment regimens: Arm A: abacavir/lamivudine 1 tablet once a day + raltegravir 400 mg (1 tablet twice a day) Arm B: abacavir/lamivudine 1 tablet once a day + ritonavir 100 mg + darunavir 800 mg once a day.

All drugs have been approved for the treatment of HIV infection. Administration: oral The study population will consist of 350 HIV-positive, HLA B5701-negative patients. At baseline, patients will be randomized 1:1 to start abacavir/lamivudine plus either raltegravir or darunavir/ritonavir. Randomization will be stratified on the basis of the screening CD4+ cell count (≤100 vs ≥100 cells/µL), to ensure balance across treatments groups 1.7 Criteria for Safety: Adverse events and laboratory assessments. 1.8 Statistical analysis: As this is a non-inferiority trial, we will calculate the difference in the proportions of patients experiencing the primary outcome in the two treatment arms and will calculate a 95% confidence interval for this. Non-inferiority of the raltegravir arm will be demonstrated if the lower limit of the 95% confidence interval is greater than -12%. In case non-inferiority will be met, analyses for superiority will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females (inpatients or outpatients) aged 18-64 years who are HIV-1 antibody seropositive, with a CD4 count <200 cells/uL.
2. All patients should be antiretroviral-naive
3. All patients should be HLA B57 or HLA B5701 negative
4. Patients must have an HIV RNA level <500,000 copies/mL
5. Patients with an active opportunistic infection could be enrolled as long as this was diagnosed more than 2 weeks prior to screening.
6. Patients must meet the following laboratory criteria. Neutrophil count > 1,000 cells/mm3 Haemoglobin > 9.0 grams/dl (men and women) Platelet count ≥ 75,000 cells/mm3 Alkaline phosphatase < 3.0 the upper limit of normal ALT and AST < 3.9 times the upper limit of normal Total bilirubin < 1.5 times the upper limit of normal.
7. Female patients of childbearing potential must be willing to use a reliable form of contraception, which will include a medically approved form of barrier contraception.
8. Patients must be able to provide written consent to comply with study requirements.

Exclusion Criteria:

1. Patients with genotypic mutations for any of the study drugs.
2. Patients with an opportunistic infection diagnosed in the 2 weeks prior to screening.
3. Female patients who are pregnant or breastfeeding.
4. Patients who are receiving any investigational drug or anti-neoplastic radiotherapy/chemotherapy other than local skin radiotherapy within 12 weeks before randomization.
5. Patients with a current history of intravenous drug abuse, alcohol or substance abuse.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
HIV RNA Viral Load | baseline and week 48
  The proportion of patients attaining an HIV RNA level <50 copies/mL after 48 weeks will be the primary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Mussini, Professor, Principal Investigator — University of Modena and ReggioEmilia
Locations (1):
- University of Modena and Reggio Emilia, Modena, Italy

IPD SHARING:
Plan to Share IPD: No